CLINICAL TRIAL: NCT03075384
Title: Application of Computer-Assisted Navigation System in the Treatment of Unilateral Complicated Zygomatic Complex Fractures: A Randomized Controlled Trial
Brief Title: Treatment of Unilateral Complicated Zygomatic Complex Fractures Using Computer-Assisted Navigation System
Status: Completed | Type: Observational
Sponsor: Xiao Zhang (Other)
Collaborators: West China College of Stomatology (Other)
Responsible Party: Sponsor-Investigator, Xiao Zhang, Principal Investigator, West China College of Stomatology
Organization: West China College of Stomatology (Other)
Other Study IDs: Xiao_owen
Record Dates: First submitted 2017-03-04; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Zygomatic Fractures
Keywords: computer-assisted navigation system
MeSH Terms: conditions — Zygomatic Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- open reduction and internal fixation: A classic method was used to treat unilateral complicated zygomatic fractures without the assistance of computer-assisted navigation system
  Interventions: Procedure: computer-assisted navigation system

INTERVENTIONS:
Procedure: computer-assisted navigation system — The computer-assisted navigation system was applied in treatment of unilateral complicated zygomatic fractures

SUMMARY:
Many studies show that computer-assisted navigation system have been available to treat zygomatic-complex fractures. However, most of them are case reports or clinical experiences lacking multiple variables and controlled design. The aim of this study was to evaluate the accuracy of the computer-assisted navigation system by a randomized controlled trial with multiple variables.

DETAILED DESCRIPTION:
In this prospective randomized controlled trial, twenty patients with unilateral complicated zygomatic fractures were divided into experimental and control groups. Patients in the experimental group were treated with open reduction and internal fixation with the assistance of surgical navigation technology, and patients in the control group without it. Preoperative and postoperative CT data were obtained to measure surgical landmarks discrepancy between the 2 groups. The Chi-square Test and t-test were conducted to test whether there was significant difference in the accuracy between the two groups. Evaluating the effect of fixation by the data and clinical symptoms.

Twenty patients with unilateral complicated zygomatic-complex fractures received operation. All patients healed and their function and facial contour were improved obviously. Postoperative clinical symptoms were not significantly different between the two groups (P>0.05). Compared with the control group, discrepancy of surgical landmarks measured by software Geomagic studio 11, Brainlabiplan CMF 3.0 were significantly low in the experimental group (P<0.05). Software measurement showed the symmetry of zygomatic area and the effect of the fixation in the experimental group were more satisfactory than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ZMC fractures including complete monofragment zygomatic or tetrapod fracture, multifragment or comminuted fracture
* Patients were sane and the age were between 18 to 60 years
* Patients suffered facial deformity and dysfunction which need be treated by operation
* There is no contraindication in patients
* The study were conducted after patient's informed consent

Exclusion Criteria:

* Cases in which technical problems or registration fails occur and patients who were lost to follow-up within 1 year are excluded from this study.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with unilateral complicated zygomatic-complex fractures
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
accuracy of the reduction of the fractures | one year

CONTACTS AND LOCATIONS:
Overall Officials: Lei Liu, DMD, Study Director — Department of Oral & Maxillofacial Surgery, West China Hospital of Stomatology, Sichuan University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Naveen Shankar A, Naveen Shankar V, Hegde N, Sharma, Prasad R. The pattern of the maxillofacial fractures - A multicentre retrospective study. J Craniomaxillofac Surg. 2012 Dec;40(8):675-9. doi: 10.1016/j.jcms.2011.11.004. Epub 2011 Dec 31. PMID 22212823
- [Background] Bogusiak K, Arkuszewski P. Characteristics and epidemiology of zygomaticomaxillary complex fractures. J Craniofac Surg. 2010 Jul;21(4):1018-23. doi: 10.1097/scs.0b013e3181e62e47. PMID 20677370
- [Background] Rana M, Warraich R, Tahir S, Iqbal A, von See C, Eckardt AM, Gellrich NC. Surgical treatment of zygomatic bone fracture using two points fixation versus three point fixation--a randomised prospective clinical trial. Trials. 2012 Apr 12;13:36. doi: 10.1186/1745-6215-13-36. PMID 22497773
- [Background] Kuhnel TS, Reichert TE. Trauma of the midface. GMS Curr Top Otorhinolaryngol Head Neck Surg. 2015 Dec 22;14:Doc06. doi: 10.3205/cto000121. eCollection 2015. PMID 26770280
- [Background] Yu H, Shen G, Wang X, Zhang S. Navigation-guided reduction and orbital floor reconstruction in the treatment of zygomatic-orbital-maxillary complex fractures. J Oral Maxillofac Surg. 2010 Jan;68(1):28-34. doi: 10.1016/j.joms.2009.07.058. PMID 20006151
- [Background] Katzen JT, Jarrahy R, Eby JB, Mathiasen RA, Margulies DR, Shahinian HK. Craniofacial and skull base trauma. J Trauma. 2003 May;54(5):1026-34. doi: 10.1097/01.TA.0000066180.14666.8B. PMID 12777923
- [Background] Jamal BT, Pfahler SM, Lane KA, Bilyk JR, Pribitkin EA, Diecidue RJ, Taub DI. Ophthalmic injuries in patients with zygomaticomaxillary complex fractures requiring surgical repair. J Oral Maxillofac Surg. 2009 May;67(5):986-9. doi: 10.1016/j.joms.2008.12.035. PMID 19375007
- [Background] Wang TH, Ma H, Tseng CS, Chou YH, Cai KL. Using Free Navigation Reference Points and Prefabricated Bone Plates for Zygoma Fracture Model Surgeries. J Med Biol Eng. 2016;36:316-324. doi: 10.1007/s40846-016-0144-x. Epub 2016 Jun 6. PMID 27441035
- [Background] Lubbers HT, Jacobsen C, Matthews F, Gratz KW, Kruse A, Obwegeser JA. Surgical navigation in craniomaxillofacial surgery: expensive toy or useful tool? A classification of different indications. J Oral Maxillofac Surg. 2011 Jan;69(1):300-8. doi: 10.1016/j.joms.2010.07.016. Epub 2010 Nov 2. No abstract available. PMID 21050633
- [Background] Westendorff C, Gulicher D, Dammann F, Reinert S, Hoffmann J. Computer-assisted surgical treatment of orbitozygomatic fractures. J Craniofac Surg. 2006 Sep;17(5):837-42. doi: 10.1097/01.scs.0000221523.80292.93. PMID 17003608
- [Background] Pham AM, Rafii AA, Metzger MC, Jamali A, Strong EB. Computer modeling and intraoperative navigation in maxillofacial surgery. Otolaryngol Head Neck Surg. 2007 Oct;137(4):624-31. doi: 10.1016/j.otohns.2007.06.719. PMID 17903581
- [Background] Morrison CS, Taylor HO, Sullivan SR. Utilization of intraoperative 3D navigation for delayed reconstruction of orbitozygomatic complex fractures. J Craniofac Surg. 2013 May;24(3):e284-6. doi: 10.1097/SCS.0b013e31828f2a71. PMID 23714993
- [Background] Scolozzi P, Terzic A. "Mirroring" computational planning, navigation guidance system, and intraoperative mobile C-arm cone-beam computed tomography with flat-panel detector: a new rationale in primary and secondary treatment of midfacial fractures? J Oral Maxillofac Surg. 2011 Jun;69(6):1697-707. doi: 10.1016/j.joms.2010.07.049. Epub 2010 Dec 24. No abstract available. PMID 21185639
- [Background] Ellis E 3rd, Kittidumkerng W. Analysis of treatment for isolated zygomaticomaxillary complex fractures. J Oral Maxillofac Surg. 1996 Apr;54(4):386-400; discussion 400-1. doi: 10.1016/s0278-2391(96)90107-x. PMID 8600255
- [Background] van Hout WM, Van Cann EM, Koole R, Rosenberg AJ. Surgical treatment of unilateral zygomaticomaxillary complex fractures: A 7-year observational study assessing treatment outcome in 153 cases. J Craniomaxillofac Surg. 2016 Nov;44(11):1859-1865. doi: 10.1016/j.jcms.2016.09.002. Epub 2016 Sep 13. PMID 27733307
- [Background] Zingg M, Laedrach K, Chen J, Chowdhury K, Vuillemin T, Sutter F, Raveh J. Classification and treatment of zygomatic fractures: a review of 1,025 cases. J Oral Maxillofac Surg. 1992 Aug;50(8):778-90. doi: 10.1016/0278-2391(92)90266-3. PMID 1634968
- [Background] Heiland M, Habermann CR, Schmelzle R. Indications and limitations of intraoperative navigation in maxillofacial surgery. J Oral Maxillofac Surg. 2004 Sep;62(9):1059-63. doi: 10.1016/j.joms.2004.02.013. PMID 15346354
- [Background] Yu H, Shen SG, Wang X, Zhang L, Zhang S. The indication and application of computer-assisted navigation in oral and maxillofacial surgery-Shanghai's experience based on 104 cases. J Craniomaxillofac Surg. 2013 Dec;41(8):770-4. doi: 10.1016/j.jcms.2013.01.016. Epub 2013 Feb 23. PMID 23462802
- [Background] Luebbers HT, Messmer P, Obwegeser JA, Zwahlen RA, Kikinis R, Graetz KW, Matthews F. Comparison of different registration methods for surgical navigation in cranio-maxillofacial surgery. J Craniomaxillofac Surg. 2008 Mar;36(2):109-16. doi: 10.1016/j.jcms.2007.09.002. Epub 2008 Feb 14. PMID 18280173
- [Background] Kang SH, Kim MK, Kim JH, Park HK, Park W. Marker-free registration for the accurate integration of CT images and the subject's anatomy during navigation surgery of the maxillary sinus. Dentomaxillofac Radiol. 2012 Dec;41(8):679-85. doi: 10.1259/dmfr/21358271. Epub 2012 Apr 12. PMID 22499127
- [Background] He Y, Zhang Y, An JG, Gong X, Feng ZQ, Guo CB. Zygomatic surface marker-assisted surgical navigation: a new computer-assisted navigation method for accurate treatment of delayed zygomatic fractures. J Oral Maxillofac Surg. 2013 Dec;71(12):2101-14. doi: 10.1016/j.joms.2013.07.003. PMID 24237774
- [Background] Zhang W, Wang C, Shen G, Wang X, Cai M, Gui H, Liu Y, Yang D. A novel device for preoperative registration and automatic tracking in cranio-maxillofacial image guided surgery. Comput Aided Surg. 2012;17(5):259-67. doi: 10.3109/10929088.2012.710251. PMID 22897358
- [Background] Fitzpatrick JM. The role of registration in accurate surgical guidance. Proc Inst Mech Eng H. 2010;224(5):607-22. doi: 10.1243/09544119JEIM589. PMID 20718266
- [Background] Jia H, Chen Q, Cao R, Yang J, Huang Q, Wang Z, Wu H. [A comparison between anatomical landmark registration and surface registration for computer-assisted endoscopic sinus surgery]. Lin Chuang Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2010 Jan;24(2):49-52, 56. Chinese. PMID 20306849
- [Background] Hardy SM, Melroy C, White DR, Dubin M, Senior B. A comparison of computer-aided surgery registration methods for endoscopic sinus surgery. Am J Rhinol. 2006 Jan-Feb;20(1):48-52. PMID 16539295